

Title: A Phase 1, Double-Blind, Parallel Group Study to Evaluate the Safety and Pharmacokinetics of Quadruple Therapy (Bismuth, Clarithromycin, and Amoxicillin) With TAK-438 Versus Quadruple Therapy With Lansoprazole.

NCT Number: NCT02892409

SAP Approve Date: 15MAY2017

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



Template Number: C-TMPL-DO-801  Version Number: 1.2 Effective Date: 14 Sep 2015

This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

# TAKEDA DEVELOPMENT CENTER STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-438\_115

A Phase 1, Double-Blind, Parallel Group Study to Evaluate the Safety and Pharmacokinetics of Quadruple Therapy (Bismuth, Clarithromycin, and Amoxicillin) With TAK-438 Versus Quadruple Therapy With Lansoprazole.

#### PHASE 1

Version: 2.0
Date: 15MAY2017

| Prepared by: |
|--------------|
| PPD |

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.




This version replaces: 1.1

**TDC Approvals:** 

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## 1.0 APPROVAL SIGNATURES

Electronic signatures can be found on the last page of this document.

**Study Title:** A Phase 1, Double-Blind, Parallel Group Study to Evaluate the Safety and

Pharmacokinetics of Quadruple Therapy (Bismuth, Clarithromycin, and

Amoxicillin) With TAK-438 Versus Quadruple Therapy With

Lansoprazole.

| PPD | Date |
|-----|------|
| | <br> |
| PPD | Date |
| PPD | Date |
| PD | Date |
| PPD | Date |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## 2.0 TABLE OF CONTENTS

| 1.0 | APPROVA | AL SIGNATURES | 2 |
|---|---|---|---|
| 2.0 | TABLE OF | F CONTENTS | 3 |
| 3.0 | LIST OF A | ABBREVIATIONS | 5 |
| 4.0 | OBJECTI\ | VES | 7 |
| | 4.1. | PRIMARY OBJECTIVES | 7 |
| | 4.2. | SECONDARY OBJECTIVES | 7 |
| | 4.3. | Additional Objectives | 7 |
| | 4.4. | STUDY DESIGN | 7 |
| 5.0 | ANALYSIS | S ENDPOINTS | 9 |
| 6.0 | DETERMI | NATION OF SAMPLE SIZE | 10 |
| 7.0 | METHODS | S OF ANALYSIS AND PRESENTATION | 11 |
| | 7.1 | GENERAL PRINCIPLES | |
| | 7.1.1 | Definitions | 11 |
| | 7.1.2 | Handling of Plasma Bismuth Concentrations at Day 14 | 11 |
| | 7.1.3 | Handling of Plasma TAK-438F/ Lansoprazole Concentrations | 13 |
| | 7.1.4 | Handling of Laboratory Test | 13 |
| | 7.1.5 | Handling of Vital Signs | 14 |
| | 7.1.6 | Handling of 12-Lead ECGs | 14 |
| | 7.1.7 | Handling of HP Breath Test | 15 |
| | 7.2 | Analysis Sets | 15 |
| | 7.3 | DISPOSITION OF SUBJECTS | 16 |
| | 7.3.1 | Study Information | 16 |
| | 7.3.2 | Screen Failures | 16 |
| | 7.3.3 | Subject Eligibility | 16 |
| | 7.3.4 | Disposition of Subjects | 17 |
| | 7.3.5 | Protocol Deviations and Analysis Sets | 17 |
| | Protoc | col Deviations | 17 |
| | Analy | sis Sets | 18 |
| | 7.4 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 18 |
| | 7.5 | MEDICAL HISTORY AND CONCURRENT MEDICAL CONDITIONS | 19 |
| | 7.6 | MEDICATION HISTORY AND CONCOMITANT MEDICATIONS | 19 |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| | 7.7 | STUDY DRUG EXPOSURE AND COMPLIANCE | 19 |
|---|---|---|---|
| | TAK-4 | 138/ Lansoprazole and Bismuth Exposure and Compliance | 19 |
| | Clarith | nromycin and Amoxicillin Exposure and Compliance | 19 |
| | 7.8 | Efficacy Analysis | 20 |
| | 7.9 | PHARMACOKINETIC ANALYSIS | |
| | Plasm | na Bismuth Concentration | 20 |
| | | na TAK-438F/ Lansoprazole Concentration | |
| | | a PK Parameters of Bismuth | |
| | | PK parameters of Bismuth | |
| | 7.10 | OTHER OUTCOMES | 21 |
| | HP Br | eath Test | |
| | 7.11 | SAFETY ANALYSIS | |
| | 7.11.1 | Adverse Events | |
| | 7.11.1 | | |
| | 7.11.1 | - | |
| | 7.11.1 | | |
| | 7.11.2 | Clinical Laboratory Evaluations | |
| | | tology and Serum Chemistry | |
| | Urinal | ysis | 25 |
| | 7.11.3 | Vital Signs | 26 |
| | 7.11.4 | 12-Lead ECGs | 26 |
| | 7.11.5 | Other Observations Related to Safety | 27 |
| | 7.12 | INTERIM ANALYSIS | 27 |
| | 7.13 | Changes in the Statistical Analysis Plan | 27 |
| 8.0 | REFEREN | CES | 28 |
| 9.0 | APPENDI | <b>(</b> | 29 |
| | 9.1 | CRITERIA FOR MARKEDLY ABNORMAL VALUES | 29 |
| | 9.1.1 | Hematology, Serum Chemistry, Vital Signs, and 12-lead ECG (except Upper MA\ Criteria of QTcF Interval) | |
| | 9.1.2 | | |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## 3.0 LIST OF ABBREVIATIONS

AE adverse event

 $Ae_{\tau}$  amount of drug excreted in urine during a dosing interval

ALT alanine aminotransferase
ALP alkaline phosphatase

AUC $_{\tau}$  area under the concentration-time curve during a dosing interval AUC $_{\infty}$  area under the plasma concentration-time curve from time 0 to infinity

AST aspartate aminotransferase

BID twice daily
BMI body mass index

CAL clarithromycin (500 mg BID), amoxicillin (1000 mg BID), and lansoprazole (30 mg

BID)

CAT clarithromycin (500 mg BID), amoxicillin (1000 mg BID), and TAK-438 (20 mg

BID)

CL/F apparent clearance after extravascular administration, calculated using the observed

value of the last quantifiable concentration

CL<sub>R</sub> renal clearance

C<sub>max</sub> maximum observed plasma concentration

CRF case report form
CV coefficient of variation
CYP cytochrome P450
ECG electrocardiogram

 $f_{e,\tau}$  Fraction of administered dose of drug excreted in urine during a dosing interval.

Molecular weight adjustment needed for metabolites.

GGT  $\gamma$ -glutamyl transferase HP  $Helicobacter\ pylori$  LDH lactate dehydrogenase LLN lower limit of normal

 $\lambda_z$  terminal disposition phase rate constant

MAV markedly abnormal values

Medical Dictionary for Regulatory Activities

PD pharmacodynamics
PK pharmacokinetics
PTE pretreatment event

QTcF QT interval corrected by Fridericia's method

SAP statistical analysis plan TAK-438F freebase of TAK-438

TEAE treatment-emergent adverse event  $t_{1/2z}$  terminal disposition phase half-life




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

 $t_{max} \hspace{2cm} time\ of\ first\ occurrence\ of\ C_{max}$ 

ULN upper limit of normal

 $V_z/F$  apparent volume of distribution during the terminal disposition phase after

extravascular administration, calculated using the observed value of the last

quantifiable concentration

WHO Drug World Health Organization Drug Dictionary




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 4.0 OBJECTIVES

#### 4.1. PRIMARY OBJECTIVES

The primary objective is to evaluate the safety, tolerability, and PK of quadruple therapy BID with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and TAK-438 (20 mg) versus quadruple therapy BID with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and lansoprazole (30 mg).

#### 4.2. SECONDARY OBJECTIVES

Not applicable

#### 4.3. ADDITIONAL OBJECTIVES

Not applicable

#### 4.4. STUDY DESIGN

This is a phase 1, double-blind, parallel group study in HP positive subjects to evaluate the safety, tolerability, and PK of quadruple therapy with bismuth, clarithromycin, amoxicillin, and TAK-438 versus quadruple therapy with bismuth, clarithromycin, amoxicillin, and lansoprazole.

Thirty HP positive male or female subjects aged 19 to 60 years, inclusive, considered eligible based on the inclusion and exclusion criteria, will participate in this study. All subjects will be enrolled and will be randomized to 1 of 2 treatment groups as indicated in Figure 1. One site in Asia will be selected to conduct this study.

The treatment phase consists of quadruple therapy BID with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and TAK-438 (20 mg) or quadruple therapy BID with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and lansoprazole (30 mg) for 14 days (Days 1 to 14). Subjects will be discharged on Day 15 after final PK blood samples are collected and all procedures performed.

Screening for potential subjects will occur between Days -28 and -2 prior to confinement at the phase 1 unit. Eligibility will be reconfirmed on Day -1. Having fasted for a minimum of 8 hours, oral doses of tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and TAK-438 (20 mg) or tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and lansoprazole (30 mg) will be administered BID from Days 1 to 14. The last dose will be on the evening of Day 14. Blood sampling for TAK-438 and lansoprazole PK measurements will be taken on Days 12 to 14 (predose evening and morning) and for bismuth PK measurements on Day 14 (pre–morning dose to 12 hours post–morning dose). Urine sampling for bismuth PK measurements will be taken on Day 14 (pre–morning dose to 12 hours post–morning dose). The subject will be confined to the phase 1 unit from Day -1 (Check-in) through to Day 15 (Check-out), and will be required to contact the study site once again for a follow-up call on Day 17 and a clinic visit on Day 42 for a HP breath test.

A schematic of the study design is included as Figure 1.

Figure 1. Schematic of Study Design




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Pretrea | tment | Treatment Period | | | Foll | ow |
|---|---|---|---|---|---|---|
| | | | | | սլ | ) |
| Screening | Check-in<br>Baseline | Confinement | | Check-<br>out | Follow-up<br>call | Follow-up<br>visit |
| Days -28<br>to -2 | Day -1 | Day 1-11 Day 12-13 Day 14 | | | Day 17 (+2<br>days) | Day 42<br>(+6 days) |
| | | Group A: CA + bismuth + lansoprazole dosing Group B: CA + bismuth + TAK-438 dosing | | | | HP breath<br>test |
| | | TAK-438 PK or<br>lansoprazole PK in<br>plasma | | | | |
| | | | Bismuth<br>PK in<br>plasma<br>and urine | | | |

Bismuth: tripotassium bismuth dicitrate (600 mg BID, equivalent to bismuth 220 mg BID); CA: clarithromycin (500 mg BID), amoxicillin (1000 mg BID); TAK-438: 20 mg BID; lansoprazole: 30 mg BID.

Blood PK samples for Bismuth: Day 14 predose (0 hours), 0.25, 0.50, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hours after morning dose.

Urine PK samples for Bismuth: Day 14 at 0 to 12 hours post-morning dose.

Blood PK samples for TAK-438 and lansoprazole: Day 12-14 predose (morning and evening)

Analyte: bismuth, TAK-438F, and lansoprazole.

Comparison of Group A and Group B:  $C_{max}$  and  $AUC_{\tau}$ .




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 5.0 ANALYSIS ENDPOINTS

- Percentage of subjects who experience at least 1 treatment-emergent adverse event (TEAE).
- Percentage of subjects who discontinue due to an adverse event (AE).
- Percentage of subjects who meet the markedly abnormal criteria for safety laboratory tests at least once postdose.
- Percentage of subjects who meet the markedly abnormal criteria for vital sign measurements at least once postdose.
- Percentage of subjects who meet the markedly abnormal criteria for safety electrocardiogram (ECG) parameters at least once postdose.
- Plasma PK parameters of tripotassium bismuth dicitrate (600 mg) when coadministered with clarithromycin (500 mg BID), amoxicillin (1000 mg BID), and TAK-438 (20 mg BID) (CAT), and coadministered with clarithromycin (500 mg BID), amoxicillin (1000 mg BID), and lansoprazole (30 mg BID) (CAL):
  - $C_{\text{max}}$  at Day 14.
  - The area under the plasma concentration-time curve during a dosing interval (AUC $_{\tau}$ ) at Day 14.
  - The amount of drug excreted in urine during a dosing interval ( $Ae_{\tau}$ ) at Day 14.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 6.0 DETERMINATION OF SAMPLE SIZE

A sample size of 30 (15 subjects per group) will be used in this exploratory study. Although this planned sample size is not primarily based on statistical considerations, it will allow precise estimation of the relative treatment effect of TAK-438 versus lansoprazole on bismuth exposure as follows:

| Estimated Ratio<br>TAK-438/Lansoprazole | CV | Expected 90% CI | Expected 95% CI |
|---|---|---|---|
| 1.5 | 0.40 | 1.15, 1.96 | 1.09, 2.07 |
| 1.5 | 0.50 | 1.07, 2.10 | 1.00, 2.25 |
| 1.5 | 0.60 | 1.00, 2.24 | 0.92, 2.44 |
| 2.0 | 0.40 | 1.53, 2.62 | 1.45, 2.76 |
| 2.0 | 0.50 | 1.43, 2.80 | 1.33, 3.00 |
| 2.0 | 0.60 | 1.34, 2.99 | 1.23, 3.25 |

CV=coefficient of variation.

These calculations allow for up to 2 dropouts per group and are based on estimates of CV of 0.40 to 0.60 for PK parameters (area under the plasma concentration-time curve from time 0 to infinity  $[AUC_{\infty}]$  and  $C_{max}$ )




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

#### 7.1 GENERAL PRINCIPLES

#### 7.1.1 Definitions

The following definitions and calculation formulas will be used.

- TEAE: An AE whose date of onset occurs on or after the start of study drug.
- PTE: An AE whose date of onset occurs before the start of study drug.
- Significant TEAE: any AEs (not including serious TEAEs) that led to an intervention, including withdrawal of drug treatment or significant additional concomitant therapy.
- Descriptive statistics: number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Study Day: The day before the first dose of the study medication will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. Other study days are defined relative to Study Day 1, e.g., the day prior to Study Day 1 is Day -1 and the day after Study Day 1 is Day 2.
- Duration of exposure to study medication (days): date of last dose of study medication date of first dose of study medication + 1
- Study drug compliance (%): (number of times "Dose Start Time" was collected) / (2\* Duration of exposure to study medication) \*100 (rounded to 1 decimal place). Study drug compliance will be calculated each group of study drugs, 1)TAK438/ lansoprazole and bismuth or 2)clarithromycin and amoxicillin.
- QTcF interval (msec): QT interval (msec) / (RR interval (msec)/1000)<sup>0.33</sup> (rounded to the nearest whole number)
- Baseline and Screening values: The last evaluable observation (i.e., non-missing) before the first dose of study medication. If no evaluable observation is obtained before the first dose, the baseline value will be missing.

## 7.1.2 Handling of Plasma Bismuth Concentrations at Day 14

For each time, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same time window, the observation with the closest sampling time to the scheduled time will be used. If there are two observations equidistant to the scheduled time, the later observation will be used.

| Time | Scheduled Time<br>From Morning Dose* at Day 14 | Time Interval (min) |
|---|---|---|
| Time | (min) | Sampling Time<br>From Morning Dose* at Day 14 |
| Pre–morning dose (0 hours) | 0 | -10 – 0 |
| 0.25 hours post–morning dose | 15 | 10 - 20 |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| 0.5 hours<br>post–morning dose | 30 | 25 - 35 |
|---------------------------------|-----|-----------|
| 0.75 hours<br>post–morning dose | 45 | 40 - 50 |
| 1.0 hour post–morning dose | 60 | 55 - 65 |
| 1.5 hours post–morning dose | 90 | 85 - 95 |
| 2.0 hours post–morning dose | 120 | 115 - 125 |
| 3.0 hours post–morning dose | 180 | 175 - 185 |
| 4.0 hours post–morning dose | 240 | 235 - 245 |
| 5.0 hours<br>post–morning dose | 300 | 295 - 305 |
| 6.0 hours post–morning dose | 360 | 355 - 365 |
| 8.0 hours post–morning dose | 480 | 470 - 490 |
| 10.0 hours<br>post–morning dose | 600 | 590 - 610 |
| 12.0 hours<br>post–morning dose | 720 | 710 - 730 |

<sup>\*</sup> Start Time of Bismuth, TAK-438, Lansoprazole at morning

Concentrations below the lower limit of quantification will be treated as zero in the analysis of concentration-time data.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## 7.1.3 Handling of Plasma TAK-438F/ Lansoprazole Concentrations

For each visit, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest sampling time to the scheduled time will be used. If there are two observations equidistant to the scheduled time, the later observation will be used.

| Visit Time | | Scheduled<br>From D | a. | Time Interval (min) |
|---|---|---|---|---|
| Visit | Time | (min) | | Sampling Time<br>From Dose* |
| Day 12 | Pre-morning dose | Morning | 0 | -10 – 0 |
| Day 12 | Pre-evening dose | Evening | 0 | -10 – 0 |
| Day 13 | Pre-morning dose | Morning | 0 | -10 – 0 |
| Day 13 | Pre-evening dose | Evening | 0 | -10 – 0 |
| Day 14 | Pre-morning dose | Morning | 0 | -10 – 0 |
| Day 14 | Pre-evening dose | Evening | 0 | -10 – 0 |

<sup>\*</sup> Start Time of Bismuth, TAK-438, Lansoprazole

Concentrations below the lower quantifiable concentration will be treated as zero in the analysis of concentration-time data.

#### 7.1.4 Handling of Laboratory Test

For each visit, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest sampling day to the scheduled study day will be used. If there are two observations equidistant to the scheduled study day, the later observation will be used.

| Visit | Scheduled Study Day | Time Interval (days) |
|----------|---------------------|----------------------|
| Visit | (days) | Study Day |
| Baseline | Study Day: -1 | -28 – -1 |
| Day 5 | Study Day: 5 | 1 – 6 |
| Day 8 | Study Day: 8 | 7 – 9 |
| Day 12 | Study Day: 12 | 10 – 12 |
| Day 13 | Study Day: 13 | 13 |
| Day 14 | Study Day: 14 | 14 |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|--------|-------------------------------|--------------------------------|
| Day 15 | Study Day: 15 | 15 |

Values below the lower limit of quantification will be handled as zero.

## 7.1.5 Handling of Vital Signs

For each visit, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest sampling time to the scheduled time will be used. If there are two observations equidistant to the scheduled time, the later observation will be used.

| Visit | Time | Scheduled Study Day | Scheduled Time<br>From Dose* | | Time Interval (min) / Study Day (days) |
|---|---|---|---|---|---|
| Visit | Time | (days) | (min) | | Assessment Time<br>From Dose* |
| Baseline | Pre-morning dose | Study Day: 1 | Morning | 0 | Study Day: -28 – 1 |
| Day 1 | Pre-evening dose | Study Day: 1 | Evening | 0 | Time: -60 – 0 |
| Day 2 to 14 | Pre-morning dose | Study Day: 2 to 14 | Morning | 0 | Time: -60 – 0 |
| Day 2 to 14 | Pre-evening dose | Study Day: 2 to 14 | Evening | 0 | Time: -60 – 0 |
| Day 15 | | Study Day: 15 | | | Study Day:<br>Post-dose – 15 |

<sup>\*</sup> Start Time of Bismuth, TAK-438, Lansoprazole

#### 7.1.6 Handling of 12-Lead ECGs

For each visit, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest sampling time to the scheduled time will be used. If there are two observations equidistant to the scheduled time, the later observation will be used.

| Visit | Time | Scheduled Study Day | Scheduled Time<br>From Dose* | Time Interval (min) / Study Day (days) |
|---|---|---|---|---|
| | Time | (days) | (min) | Assessment Time<br>From Dose* |
| Baseline | Pre-morning dose | Study Day: 1 | Morning 0 | Study Day: -28 – 1 |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Visit | Time | Scheduled Study Day (days) Scheduled Time From Dose* | | Time Interval (min) / Study Day (days) Assessment Time | |
|---|---|---|---|---|---|
| | | , J, | (min) | | From Dose* |
| Day 3 | Pre-morning dose | Study Day: 3 | Morning | 0 | Time: -60 – 0 |
| Day 7 | Pre-morning dose | Study Day: 7 | Morning | 0 | Time: -60 – 0 |
| | Pre-morning dose | | Morning | 0 | Time: -60 – 0 |
| | 1 hour post-<br>morning<br>dose | | Morning | 60 | Time: 0< – 90 |
| Day 14 | 2 hours post-<br>morning<br>dose | Study Day: 14 | | Time: 90< – 180 | |
| | 4 hours post-<br>morning<br>dose | | Morning | 240 | Time: 180< – 300 |
| Day 15 | | Study Day: 15 | | | Study Day:<br>Post-dose – 15 |

<sup>\*</sup> Start Time of Bismuth, TAK-438, Lansoprazole

## 7.1.7 Handling of HP Breath Test

For each visit, all evaluable observation (i.e., non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest sampling day to the scheduled study day will be used. If there are two observations equidistant to the scheduled study day, the later observation will be used.

| Visit | Scheduled Study Day | Time Interval (days) |
|-----------|---------------------|----------------------|
| VISIt | (days) | Study Day |
| Screening | -2 | -28 – -2 |
| Day 42 | 42 | Post-dose – 48 |

#### 7.2 ANALYSIS SETS

The safety analysis set used for primary analysis will consist of subjects who received at least 1 dose of the study drug.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

The PK analysis set will consist of subjects who received the study drug, who have sufficient plasma/urine concentration data to calculate at least 1 pharmacokinetic parameter, and completed the minimum protocol specified procedures with no significant protocol deviations listed below:

- Subjects who did not meet inclusion criteria #3, #4 or #5

- Subjects who met exclusion criteria #1, #4, #6, #7, #8, #10, #11, #13, #14, #15, #16, #17, #21, or #22
- Subjects who have violated the rules specified in section 7.3 (excluded medications and dietary products) of the protocol up to end of Day 14
- Subjects with study medication compliance of less than 100%

#### 7.3 DISPOSITION OF SUBJECTS

#### 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form
Analysis Variables: Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods: (1) Study Information

Study information shown in the analysis variables section will be provided.

#### 7.3.2 Screen Failures

Analysis Set: All Subjects Who Were Not Randomized

Analysis Variables: Age (years)  $[Min \le -30, 30 \le -50, 50 \le -50, 50 \le -50]$ 

Gender [Male, Female]

Race [American Indian or Alaska Native, Asian, Black or African American,

Native Hawaiian or Other Pacific Islander, White]

Analytical Methods: (1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided.

#### 7.3.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Variables: Eligibility Status [Yes, No]

Primary Reason for Subject Not Being Eligible [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up, Voluntary Withdrawal,




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

Study Termination,

Did Not Meet Entrance Criteria,

Other]

Analytical Methods: (1) Eligibility for Randomization

Frequency distributions will be provided. When calculating the percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will

be used as the denominator.

7.3.4 Disposition of Subjects

Analysis Set: Randomized Set

Analysis Variables: Study Drug Administration Status [No]

Reason for Not Being Treated [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Pregnancy, Other]

Study Drug Completion Status [Completed Study Drug,

Prematurely Discontinued Study Drug]

Reason for Discontinuation of Study Drug [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Pregnancy, Other]

Analytical Methods: (1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of study drug, the total number of subjects

who prematurely discontinued the study drug will be used as the denominator.

#### 7.3.5 Protocol Deviations and Analysis Sets

#### **Protocol Deviations**

Analysis Set: Randomized Set

Analysis Variables: Protocol Deviation [Entry Criteria, Concomitant Medication,

Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria

Analytical Methods: (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## **Analysis Sets**

Analysis Set: Randomized Set Analysis Variables: Analysis Sets

> PK Analysis Set [Included] Safety Analysis Set [Included]

Analytical Methods: (1) Analysis Sets

Frequency distributions will be provided by treatment group and overall.

#### 7.4 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Analysis Set: PK Analysis Set

Safety Analysis Set

Analysis Variables: Age (years)  $[Min \le - <30, 30 \le - <50, 50 \le - <=Max]$ 

Gender [Male, Female]

Race [American Indian or Alaska Native, Asian,

Black or African American,

Native Hawaiian or Other Pacific Islander,

White]

Height (cm) [Min<= - <150, 150<= - <160,

 $160 \le -170, 170 \le -180$ 

Weight (kg) (Baseline) [Min<= - <50.0, 50.0<= - <60.0,

60.0<= - <70.0, 70.0<= - <80.0,

 $80.0 \le - \le Max$ 

BMI  $(kg/m^2)$  (Baseline) [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le - \le Max$ 

Smoking Classification [The Subject Has Never Smoked,

The Subject Is a Current Smoker,

The Subject Is an Ex-smoker]

Consumption of Alcohol [Drink Every day,

Drink a Couple of Days Per Week, Drink a Couple of Days Per Month,

Never Drink]

Consumption of Caffeine [Yes, No]

CYP2C19 Genotype [\*1/\*1, \*1/\*2, \*1/\*3, \*2/\*2, \*2/\*3, \*3/\*3]

#### Analytical Methods: (1) Summary of Demographics and Other Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided by treatment group and overall.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 7.5 MEDICAL HISTORY AND CONCURRENT MEDICAL CONDITIONS

Medical history is defined as significant conditions or diseases that stopped at or prior to the time of informed consent. Concurrent medical conditions are defined as significant conditions ongoing or present at the time of informed consent.

Medical history and concurrent medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 19.0 or higher) coding system.

There will be no analysis of medical history and concurrent medical conditions.

#### 7.6 MEDICATION HISTORY AND CONCOMITANT MEDICATIONS

Medication history information includes any medication relevant to eligibility criteria stopped prior to signing of informed consent. Concomitant medications are recorded on the eCRF and include any medications, other than the study drug, taken at any time between informed consent and on or prior to the last dose of study drug.

Medication history and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO Drug) version 2016Q1 or higher.

There will be no analysis of medication history and concomitant medications.

#### 7.7 STUDY DRUG EXPOSURE AND COMPLIANCE

## TAK-438/ Lansoprazole and Bismuth Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis Variables: Duration of Exposure to Study Drug (days)

Study Drug Compliance (%) [Min<= - <50.0, 50.0<= - <70.0, 70.0<= -

<90.0, 90.0<= - <=Max]

Analytical Methods: (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided by treatment group and overall.

#### Clarithromycin and Amoxicillin Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis Variables: Duration of Exposure to Study Drug (days)

Study Drug Compliance (%) [Min<= - <50.0, 50.0<= - <70.0, 70.0<= -

<90.0, 90.0 <= - <= Max

Analytical Methods: (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided by treatment group and overall.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 7.8 EFFICACY ANALYSIS

Not applicable.

#### 7.9 PHARMACOKINETIC ANALYSIS

#### Plasma Bismuth Concentration

Analysis Set: PK Analysis Set

Analysis Variable: Plasma Bismuth Concentrations

Time Point: Pre-morning dose (0 hours) and 0.25, 0.50, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0,

12.0 hours post-morning dose during Day 14

Analytical Methods: Following analysis will be provided by treatment group.

(1) Summary of Plasma Concentrations by Time Point

Descriptive statistics for observed values will be provided for each time point. In

addition, geometric mean, and %CV will be provided

(2) Concentration-time Profiles of Bismuth for Individual Subjects

Observed values will be plotted using individual case plot.

(3) Mean Concentration-time Profiles with Standard Deviations

Mean of plasma concentration will be plotted by time point using linear scale and

natural log scale.

#### Plasma TAK-438F/ Lansoprazole Concentration

Analysis Set: PK Analysis Set

Analysis Variable: Plasma TAK-438F Concentrations

Plasma Lansoprazole Concentrations

Visit and Time Point: Day 12 Pre-morning dose, Day 12 Pre-evening dose, Day 13 Pre-morning dose, Day 13

Pre-evening dose, Day 14 Pre-morning dose and Day 14 Pre-evening dose

Analytical Methods: (1) Summary of Plasma Concentrations by Time Point

Descriptive statistics for observed values will be provided for each visit and time point.

In addition, geometric mean, and %CV will be provided.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### Plasma PK Parameters of Bismuth

Analysis Set: PK Analysis Set

Analysis Variable: Plasma PK Parameters of Bismuth

 $\begin{array}{ccc} C_{max} & AUC_{\tau} & CL/F \\ \lambda_{z} & t_{1/2z} & t_{max} \end{array}$ 

 $V_z/F$ 

Visit Day 14

Analytical Methods: For all variables, Summary (1) will be provided by treatment group.

For  $C_{max}$  and  $AUC_{\tau}$ , Summary (2) will be provided.

(1) Summary of Plasma PK Parameters

Descriptive statistics for PK parameters will be provided. In addition, geometric mean and %CV will be computed for  $C_{max}$  and  $AUC_{\tau}$ .

(2) Analysis of Variance with Natural log-transformed  $AUC_{\tau}$  and  $C_{max}$ 

Two-sided confidence intervals (90% and 95% confidence level) of the ratio between administration conditions (bismuth with CAL and bismuth with CAT) will be calculated using an analysis of variance with natural log-transformed  $AUC_{\tau}$  and  $C_{max}$  of bismuth.

#### Urine PK parameters of Bismuth

Analysis Set: PK Analysis Set

Analysis Variable: Urine PK parameters of Bismuth

 $Ae_{\tau}$   $f_{e,\,\tau}$   $CL_R$ 

Visit Day 14

Analytical Methods: (1) Summary of Urine PK Parameters

Descriptive statistics for PK parameters will be provided.

#### 7.10 OTHER OUTCOMES

#### **HP Breath Test**

Analysis Set: Safety Analysis Set
Analysis Variable: HP Breath Test

Visit Screening and Day 42

Analytical Methods: (1) Summary of HP Breath Test

Frequency distributions will be provided by treatment group and overall.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 7.11 SAFETY ANALYSIS

#### 7.11.1 Adverse Events

#### 7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: TEAE

Categories: Relationship to Study Drug

Relationship to TAK-438/ [Related, Not Related]

Lansoprazole

Relationship to Bismuth
Relationship to Clarithromycin
Relationship to Amoxicillin
Intensity

[Related, Not Related]
[Related, Not Related]
[Related, Not Related]
[Related, Not Related]

Analytical Methods: The following summaries will be provided for each treatment group.

#### (1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 6) Relationship of Serious Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 7) Serious Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 8) Treatment-Emergent Adverse Events Resulting in Death (number of events, number and percentage of subjects)
- 9) Significant Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 10) Relationship of Significant Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

#### Number of subjects

• Summaries for 2), 6) and 10)

A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.

• Summary for 3)




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), 6) and 10)

A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated.

#### 7.11.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: TEAE

Categories: Intensity [Mild, Moderate, Severe]

Analytical Methods: The following summaries will be provided using frequency distribution for each treatment

group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by SOC only or PT only.

Drug-related TEAEs will be summarized for TAK-438/ Lansoprazole, Bismuth, Clarithromycin and Amoxicillin, respectively.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (10) Drug-Related Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

• Summary tables other than (5), and (6)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

#### 7.11.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Variables: PTE

Analytical Methods: The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will

be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in

that PT.

#### 7.11.2 Clinical Laboratory Evaluations

#### Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

Analysis Variables: Hematology

RBCs ( $\times 10^{12}$ /L) WBCs ( $\times 10^{9}$ /L) Hemoglobin (g/L)

Hematocrit (%) Platelets  $(\times 10^9/L)$ 

White Blood Cell Fractions (Neutrophils (%), Eosinophils (%), Basophils (%),

Monocytes (%), Lymphocytes (%))

PT/INR aPTT (sec) Reticulocyte count ( $\times 10^9/L$ )

Serum Chemistry

ALT (U/L) Alkaline phosphatase (U/L) AST (U/L)

GGT (U/L) Total Bilirubin (µmol/L) LDH (U/L)

Creatine kinase (U/L) Creatine kinase MB (µg/L) Albumin (g/L)




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

Total Protein (g/L) Serum creatinine (umol/L) Blood urea nitrogen (mmol/L)

Uric Acid (mmol/L) HDL Cholesterol (mmol/L) LDL Cholesterol (mmol/L)

Triglycerides (mmol/L) Glucose (mmol/L) Potassium (mmol/L)
Sodium (mmol/L) Magnesium (mmol/L) Calcium (mmol/L)

Chloride (mmol/L) Amylase (U/L)

Visit: Baseline, Day 5, 8, 12, 13, 14, 15

Analytical Methods: The following summaries will be provided for each treatment group.

## (1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - baseline) will be provided for each visit.

#### (2) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided. For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### (3) Number and Percentage of Subjects with Markedly Abnormal Values of Laboratory Test results

Overall frequency distributions of MAV during treatment phase will be provided. If a laboratory test result has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### Urinalysis

Analysis Set: Safety Analysis Set

Analysis Variables : pH  $[Min \le -<5.0, 5.0 \le -<=8.5, 8.5 < -<=Max]$ 

Specific gravity [Min<= - <1.005, 1.005<= - <=1.030, 1.030< - <=Max]

Protein [Negative, Positive] Glucose [Negative, Positive] **Nitrites** [Negative, Positive] Bilirubin [Negative, Positive] Hemoglobin [Negative, Positive] Ketones [Negative, Positive] Leucocytes [Negative, Positive] Urobilinogen [Negative, Positive]

Visit: Baseline, Day 5, 8, 12, 13, 14, 15

Analytical Methods: The following summaries will be provided for each treatment group.

(1) Summary of Shifts of Urine Laboratory Test Results




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

7.11.3 Vital Signs

Analysis Set: Safety Analysis Set Analysis Variables: Body Temperature (°C)

> Systolic Blood Pressure (mmHg) Diastolic Blood Pressure (mmHg)

Respiratory Rate (bpm)

Pulse (bpm)

Visit: Baseline, Day 1at Pre–evening dose, Day 2 to 14 at Pre–morning dose, Day 2 to 14 Pre–

evening dose, , Day 15

Analytical Methods: For each variable, following summary will be provided by treatment group.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit – baseline) will be provided for each visit.

(2) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters

Overall frequency distributions of MAV during treatment phase will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### 7.11.4 12-Lead ECGs

Analysis Set: Safety Analysis Set Analysis Variables: Heart Rate (bpm)

RR Interval (msec)
PR Interval (msec)
QT Interval (msec)
QTcF Interval (msec)
QRS Interval (msec)

12-Lead ECG Interpretation ["Within Normal Limits",

"Abnormal, Not Clinically Significant",
"Abnormal, Clinically Significant"]

Visit: Baseline, Day 3, Day 7 at Pre–morning dose, Day 14 at Pre–morning dose, 1, 2, 4 hour Post–

morning dose, Day 15

Analytical Methods: For each variable other than 12-lead ECG interpretations, summary (1) will be provided by

treatment group.

For 12-lead ECG interpretations, summary (3) will be provided by treatment group.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### (1) Summary of ECG Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit – baseline) will be provided for each visit.

## (2) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters

Overall frequency distributions of MAV during treatment phase will be provided. If an ECG parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### (3) Summary of Shifts of ECG Parameters

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.11.5 Other Observations Related to Safety

Not applicable

#### 7.12 INTERIM ANALYSIS

Not applicable

#### 7.13 CHANGES IN THE STATISTICAL ANALYSIS PLAN

Time intervals in 7.1.5 and 7.1.6 were modified from SAP version 1.0 to include all records for premorning dose, pre-evening dose, and Day 15 as well as to correct misspecification for post-morning dose.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

## 8.0 REFERENCES

Not applicable




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### 9.0 APPENDIX

#### 9.1 CRITERIA FOR MARKEDLY ABNORMAL VALUES

9.1.1 Hematology, Serum Chemistry, Vital Signs, and 12-lead ECG (except Upper MAV Criteria of QTcF Interval)

For each parameter, all evaluable data (i.e., non-missing data) obtained up to Day 15 will be classified as a MAV or not. The criteria in the table below will be used.

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

Hematology

| Parameter | MAV Criteria | |
|-------------------------------|----------------|----------------|
| | Lower Criteria | Upper Criteria |
| $RBCs (\times 10^{12}/L)$ | <0.8×LLN | >1.2×ULN |
| WBCs ( $\times 10^9$ /L) | <0.5×LLN | >1.5×ULN |
| Hemoglobin (g/L) | <0.8×LLN | >1.2×ULN |
| Hematocrit (%) | <0.8×LLN | >1.2×ULN |
| Platelets ( $\times 10^9/L$ ) | <75 | >600 |
| Neutrophils (%) | <0.5×LLN | >1.5×ULN |
| Eosinophils (%) | - | >2×ULN |
| Basophils (%) | - | >3×ULN |
| Monocytes (%) | - | >2×ULN |
| Lymphocytes (%) | <0.5×LLN | >1.5×ULN |
| aPTT (sec) | | >1.5×ULN |
| PT/INR | | >1.5 |

**Serum Chemistry** 

| Parameter | MAV Criteria | |
|----------------------------|----------------|----------------|
| Farameter | Lower Criteria | Upper Criteria |
| ALT (U/L) | - | >3×ULN |
| Alkaline phosphatase (U/L) | - | >3×ULN |
| AST (U/L) | - | >3×ULN |
| GGT (U/L) | - | >3×ULN |
| Total Bilirubin (µmol/L) | - | >34.2 |
| Creatine kinase (U/L) | - | >5×ULN |
| Albumin (g/L) | <25 | - |




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Parameter | MAV Criteria | |
|------------------------------|----------------|----------------|
| Faranictei | Lower Criteria | Upper Criteria |
| Total Protein (g/L) | <0.8×LLN | >1.2×ULN |
| Blood urea nitrogen (mmol/L) | - | >10.7 |
| Uric acid (mmol/L) | - | >0.773 |
| Triglycerides (mmol/L) | - | >2.5×ULN |
| Glucose (mmol/L) | <2.8 | >19.4 |
| Potassium (mmol/L) | <3.0 | >6.0 |
| Sodium (mmol/L) | <130 | >150 |
| Magnesium (mmol/L) | <0.5 | >1.2 |
| Calcium (mmol/L) | <1.75 | >2.88 |
| Chloride (mmol/L) | <75 | >126 |
| Amylase (U/L) | - | >2×ULN |
| Serum creatinine (µmol/L) | - | >177 |

#### **Vital Signs**

| Parameter | MAV Criteria | |
|---------------------------------|----------------|----------------|
| Faraniciei | Lower Criteria | Upper Criteria |
| Body Temperature (°C) | <35.6 | >37.7 |
| Systolic Blood Pressure (mmHg) | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | <50 | >110 |
| Pulse (bpm) | <50 | >120 |

#### 12-lead ECG

| Parameter | MAV Criteria | |
|----------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | <50 | >120 |
| QT Interval (msec) | <=50 | >=460 |
| QTcF Interval (msec) | <=50 | - |

#### 9.1.2 12-lead ECG (Upper MAV Criteria of QTcF Interval)

All evaluable data (i.e., non-missing data) obtained up to Day 15 will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
  - Observed value is less than 450 msec and not missing.
  - Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.




This version replaces: 1.1

Parent Document: C-SOP-DO-800

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Parameter | MAV Criteria | |
|---|---|---|
| Farameter | Lower Criteria | Upper Criteria |
| QTcF Interval (msec) | - | If either of the following conditions is met: • observed value >=500 • change from baseline >= 30 and observed value >=450 |

## Statistical Analysis Plan

## ELECTRONIC SIGNATURES

| EEE THO WE STOT WITCHES | | |
|---|---|---|
| Signed by | Meaning of Signatur | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
| PPD | Clinical Pharmacology Approval | 17-May-2017 08:17 UTC |
| | Pharmacovigilance Approval | 17-May-2017 13:37 UTC |
| | Clinical Science Approval | 18-May-2017 00:51 UTC |
| | Biostatistics Approval | 19-May-2017 08:39 UTC |
| | Biostatistics Approval | 22-May-2017 01:59 UTC |
| | Clinical Science Approval Biostatistics Approval | 18-May-2017 00:51 UTC<br>19-May-2017 08:39 UTC |